CLINICAL TRIAL: NCT05665088
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Efficacy and Safety Study of PRN Dosing of BXCL501 Over a 12 Week Treatment Period in Subjects With Agitation Associated With Dementia
Brief Title: Dexmedetomidine in the Treatment of Agitation Associated With Dementia (TRANQUILITY III)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated for business reasons; not due to safety or efficacy concerns
Sponsor: BioXcel Therapeutics Inc (Industry)
Collaborators: Cognitive Research Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BXCL501-304
Record Dates: First submitted 2022-12-16; First posted 2022-12-27 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Agitation; Dementia
MeSH Terms: conditions — Psychomotor Agitation; Dementia | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double-Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1- 40 Micrograms (Experimental): Sublingual film containing 40 Micrograms Dexmedetomidine
  Interventions: Drug: BXCL501
- Cohort 2- 60 Micrograms (Experimental): Sublingual film containing 60 Micrograms Dexmedetomidine
  Interventions: Drug: BXCL501
- Placebo (Placebo Comparator): Sublingual Placebo film
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: BXCL501 — Sublingual Film
  Other Names: Dexmedetomidine
  Arms: Cohort 1- 40 Micrograms; Cohort 2- 60 Micrograms
Drug: Matching Placebo — Sublingual Placebo Film
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
A study to determine the safety and efficacy of BXCL501 dosing for episodes of agitation associated with dementia when they occur (given as needed [PRN]), for a maximum of 168 doses within a 12-week treatment period.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled, parallel group, 3-arm study assessing efficacy, safety, and tolerability of two doses of BXCL501 in male and female subjects (65 years and older) with acute psychomotor agitation associated with dementia.

Approximately 150 subjects will participate in this study. Subjects will receive a single film consisting of BXCL501 40 µg dose or BXCL501 60 µg dose or placebo. Subjects must reside in a care facility where all study-related procedures and study drug dosing will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects must have a diagnosis of probable Alzheimer's disease based on NIA-AA criteria (2018). If subject biomarker data are unavailable, per the 2018 NIA-AA diagnostic criteria, the clinical diagnosis of probable AD will be based on the 2011 NIA-AA criteria
2. Episodes of psychomotor agitation (e.g., kick, bite, flailing)
3. Subjects exhibit behaviors that are congruent with the International Psychogeriatric Association criterion for agitation representing a change from the subject's usual behavior
4. A score of 0 to 20 on the Mini-Mental State Exam (MMSE) and require moderate to full assistance with activities of daily living
5. Subjects who read, understand, and provide written informed consent, or who have a LAR to provide consent on their behalf
6. Subjects who are deemed to be medically appropriate for study participation by the principal investigator
7. Participants who agree to use a medically acceptable and effective birth control method

Exclusion Criteria:

1. Subjects with dementia or other memory impairment not due to probable AD.
2. Clinical diagnosis of probable AD should not be applied when there is evidence of a cerebrovascular incident temporally related to the worsening of cognitive function.
3. Subjects with agitation caused by acute intoxication.
4. Subjects with significant risk of suicide or homicide per the investigator's assessment.
5. Subjects who are medically unstable or in recovery. Note: Subjects with a remote (>5 years) history of stroke may be included, regardless of size/location.
6. History of clinically significant syncope or syncopal attacks, orthostatic hypotension within the past 2 years, current evidence of hypovolemia, orthostatic hypotension, bradycardia.
7. Subjects with laboratory or ECG abnormalities.
8. Subjects who have received an investigational drug within 30 days prior to Screening.
9. Subjects who are currently suffering from substance abuse.
10. Subjects with a potential cause for delirium (relatively recent onset agitation and dementia)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Positive and Negative Syndrome Scale- Excited Component (PEC) total score | 120 minutes post-dose for first episode of agitation
  The Positive and Negative Syndrome Scale - Excited Component (PEC) comprises 5 items associated with agitation: poor impulse control, tension, hostility, uncooperativeness, and excitement; each scored 1 (minimum) to 7 (maximum). The PEC, the sum of these 5 subscales, thus ranges from 5 (absence of agitation) to 35 (extremely severe)

SECONDARY OUTCOMES:
Change from baseline in Positive and Negative Syndrome Scale- Excited Component (PEC) total score | 60 minutes post-dose for first episode of agitation
  The Positive and Negative Syndrome Scale - Excited Component (PEC) comprises 5 items associated with agitation: poor impulse control, tension, hostility, uncooperativeness, and excitement; each scored 1 (minimum) to 7 (maximum). The PEC, the sum of these 5 subscales, thus ranges from 5 (absence of agitation) to 35 (extremely severe)
Change from baseline in Positive and Negative Syndrome Scale- Excited Component (PEC) total score | 30 minutes post-dose for first episode of agitation
  The Positive and Negative Syndrome Scale - Excited Component (PEC) comprises 5 items associated with agitation: poor impulse control, tension, hostility, uncooperativeness, and excitement; each scored 1 (minimum) to 7 (maximum). The PEC, the sum of these 5 subscales, thus ranges from 5 (absence of agitation) to 35 (extremely severe)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Risinger, MD, Study Chair — BioXcel Therapeutics
Locations (7):
- United States (7):
  - BioXcel Clinical Research Site, Los Alamitos, California
  - BioXcel Clinical Research Site, Daytona Beach, Florida
  - BioXcel Clinical Research Site, Maitland, Florida
  - BioXcel Clinical Research Site, The Villages, Florida
  - BioXcel Clinical Research Site, Marrero, Louisiana
  - BioXcel Clinical Research Site, Springfield, Massachusetts
  - BioXcel Clinical Research Site, Toms River, New Jersey

IPD SHARING:
Plan to Share IPD: No